CLINICAL TRIAL: NCT02976129
Title: Phase 2 Study to Investigate the Efficacy, Safety, and Tolerability of Six Weeks Treatment With V565 in Subjects With Active Crohn's Disease
Brief Title: A Six Week Efficacy, Safety and Tolerability Study of V565 in Crohn's Disease
Acronym: HarbOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VHsquared Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V56502
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- V565 (Experimental): V565 three times a day (TID) PO for 6 weeks
  Interventions: Drug: V565
- Placebo (Placebo Comparator): Placebo TID PO for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: V565 — Daily dosing of V565 three times a day orally for 6 weeks
  Arms: V565
Drug: Placebo — Daily dosing of placebo three times a day orally for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of V565 in participants with active Crohn's Disease (CD).

DETAILED DESCRIPTION:
This study will be a multiple-site, double-blind, placebo-controlled, parallel-group study in approximately 126 subjects with a confirmed diagnosis of CD for at least three months and have CD involving the ileum and/or colon. Following a screening period of up to 28 days, subjects will be randomly allocated into one of two treatment arms: either V565 or placebo using a 2:1 active:placebo ratio for a treatment period of 6 weeks.

Subjects will be treated with study drug as an add-on to any permitted stable medications already being taken for CD.

ELIGIBILITY:
Inclusion Criteria:

* History of Crohn's Disease of at least 3 months duration prior to screening
* Crohn's Disease Activity Index (CDAI) score of ≥220 to ≤450 during screening
* C-reactive protein (CRP) ≥5 mg/L (or, if CRP is normal, faecal calprotectin (FCP) ≥250 µg/g) at screening
* Permitted CD medication regimen expected to remain stable during the period of the study

Exclusion Criteria:

* Previous lack of response or current contra-indication to an anti-tumour necrosis factor α (anti-TNFα) agent
* Certain complications of Crohn's Disease that would make it hard to assess response to study drug
* Known history or suspicion of inflammatory bowel disease other than Crohn's disease
* History of tuberculosis (TB) or latent TB infection that has not been treated
* Any significant illness or condition which would preclude effective participation in the study
* GI infection as demonstrated by presence of enteric pathogens
* Pregnant or lactating women
* Abdominal surgery in the previous 6 months
* Unsuitable for inclusion in the study in the opinion of the investigator or sponsor for any reason that may compromise the subject's safety or confound data interpretation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-12; Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Nurbhai, MBChB MRCP, Study Director — VHsquared Ltd.
Locations (94):
- United States (6):
  - Advanced Research Center, Inc., Anaheim, California
  - West Central Gastroenterology, Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Galiz Research, LLC, Miami Springs, Florida
  - Northwestern University, Evanston, Illinois
  - Clinical Trials of America, Mount Airy, North Carolina
- Austria (4):
  - Klinikum Klagenfurt am Wörtersee, Klagenfurt
  - LKH - Universitatsklinikum, Salzburg
  - AKH - Medizinische Universität Wien, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Canada (3):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Science Centre, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
- Czechia (5):
  - Vojenska nemocnice Brno, Brno
  - Nemocnice Horovice, Hořovice
  - Hepato-Gastroenterologie HK, Hradec Králové
  - Poliklinika MEDICINA PLUS, Prague
  - Mediendo s.r.o., Prague
- Germany (14):
  - Praxiszentrum Alte Maelzerei, Regensburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Carl Gustav Carus TU, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig
  - Charite Universitaetsmedizin, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Staedisches Klinikum, Brandenburg
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Studiengesellschaft BSF, Halle
  - Hamburgisches Forschungsinstitut fuer CED, Hamburg
  - Asklepios Klinik Hamburg, Hamburg
  - Praxis fuer Magen, Heidelberg
  - EUGASTRO GmbH, Leipzig
  - Klinik u Poliklinik f Gastro, Leipzig
- Hungary (7):
  - DRC Gyogyszervizsgalo, Balatonfüred
  - Obudai Egeszsegugyi, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Endomedix Diagnosztikai, Budapest
  - Petz Aladar Hospital, Győr
  - Clinfan Szolgaltato Kft., Szekszárd
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Maastricht University Medical Center, Maastricht
- Norway (2):
  - Akershus universitetssykehus HF, Lørenskog
  - Universitetssykehuset Nord-Norge, Tromsø
- Poland (9):
  - Polimedica Centrum Badan, Profilaktyki I Leczenia, Kielce
  - Indywidualna Specjalistyczna, Knurów
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - SOLUMED Centrum Medyczne, Poznan
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Specjalistyczna Praktyka, Sopot
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Clinical Health Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Zemun, Belgrade
  - Clinical Center Nis, Niš
- Slovakia (8):
  - Alian s.r.o, Bardejov
  - Uni nemocnica Bratislava, Bratislava
  - Nemocnica A.Lena Humenne, n.o, Humenné
  - Nemocnica s poliklinikou S. Kukuru Michalovce, a.s, Michalovce
  - KM Management spol. s r.o., Nitra
  - Gastromedic, s.r.o, Nové Zámky
  - Gastro I, s.r.o., Prešov
  - Svet zdravia a.s., Rimavská Sobota
- Ukraine (21):
  - Brovary Central District Hospital, Brovary
  - Chernivtsi RCH Dep of Surgery HSEI of Ukr Bukovinian SMU, Chernivtsi
  - Limited Liability Company Medical Center Family Medicine Clinic, Dnipro
  - Hospital for War Veterans, Kharkiv
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - Municipal Institution of Public Health Kharkiv City Clinic #9, Kharkiv
  - CI of Healthcare Kharkiv Reg Clin Hospital, Kharkiv
  - CI Ye.Ye.Karabelesh Kherson City Clinical Hosp, Kherson
  - PPC Atsynus, Kirovohrad
  - LLC Treatment and Diagnostic Center Adonis Plus, Kyiv
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv
  - Medical Centre CONSILIUM MEDICAL, Kyiv
  - Lviv Clinical Hospital at Railway Transport of Division Healthcare Center PJSC, Lviv
  - Lviv Regional Clinical Hospital, Lviv
  - CI Sumy City Clinical Hospital #1 Dept of Therapy Sumy SU Med Inst, Sumy
  - CI of SRC Sumy RCH Dept of Gastroenterology Sumy SU MI, Sumy
  - Medical Center Pulse, Vinnytsia
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia M.I.Pyrogov Regional Clinical Hospital, Vinnytsia
  - CI City Clinical Hospital #6, Zaporizhzhia
  - CI City Hospital #1, Zaporizhzhia
- United Kingdom (8):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Whipps Cross University Hospital, Leytonstone, London
  - St Mark's Hospital, Harrow, Middlesex
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Queen Elizabeth University Hospital, Glasgow, Strathclyde
  - Neath Port Talbot Hospital, Swansea, West Glamorgan
  - St Thomas' Hospital, London

RESULTS

PARTICIPANT FLOW:
Groups:
- V565: V565 three times daily (TID) PO for 6 weeks
  V565: Daily dosing of V565 three times a day orally for 6 weeks
- Placebo: Placebo three times daily (TID) PO for 6 weeks
  Placebo: Daily dosing of placebo three times a day orally for 6 weeks
Period: Overall Study
Arm/Group | V565 | Placebo
Started | 82 | 43
Completed | 77 | 41
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- V565: V565 TID PO for 6 weeks
  V565: Daily dosing of V565 three times a day orally for 6 weeks
- Total: Total of all reporting groups
Arm/Group | V565 | Placebo | Total
Number analyzed (Participants) | 82 | 43 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (14.05) | 37.2 (12.08) | 37.5 (13.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 19 | 51
  Male | 50 | 24 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 82 | 39 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Hungary | 4 | 1 | 5
  United States | 4 | 3 | 7
  Czechia | 18 | 11 | 29
  Ukraine | 22 | 12 | 34
  United Kingdom | 4 | 5 | 9
  Canada | 1 | 1 | 2
  Austria | 3 | 0 | 3
  Netherlands | 1 | 0 | 1
  Norway | 1 | 0 | 1
  Poland | 9 | 5 | 14
  Slovakia | 6 | 2 | 8
  Serbia | 5 | 1 | 6
  Germany | 4 | 2 | 6
Baseline Crohn's Disease Activity Index [Mean (Standard Deviation); unit: units on a scale] — Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450
  units on a scale | 316.34 (71.283) | 296.69 (64.334) | 309.69 (69.379)
Baseline C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] — Baseline level of C-Reactive Protein (CRP) for those subjects qualifying for the study based on CRP Population: Subjects were recruited into the study if their baseline CRP value was greater than or equal to 5mg/L OR if their baseline faecal calprotectin (FCP) measure was greater than or equal to 250µg/g. Data are reported for only those patients whose baseline CRP was greater than or equal to 5mg/L
  mg/L
    number analyzed (Participants) | 59 | 33 | 92
    (all) | 59 (21.9) | 18.7 (14.56) | 20.8 (17.13)
Baseline Faecal Calprotectin (FCP) [Mean (Standard Deviation); unit: µg/g] — Baseline Faecal Calprotectin (FCP) level for those subjects qualifying for the study on FCP Population: Subjects were recruited into the study if their baseline CRP value was greater than or equal to 5mg/L OR if their baseline FCP measure was greater than or equal to 250µg/g. Data are reported for only those patients whose baseline FCP was greater than or equal to 250µg/g
  µg/g
    number analyzed (Participants) | 23 | 10 | 33
    (all) | 1082.619 (804.2154) | 1091.217 (974.0855) | 1085.224 (843.5207)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Response to Therapy, Defined as Reduction in the CDAI Score and in Inflammatory Markers CRP or FCP at Day 42.
Description: Number of responders at Day 42, defined as subjects achieving both CDAI ≥ 70-point reduction from baseline or CDAI score < 150, and a reduction of ≥ 40% from the baseline value of CRP or FCP.
  Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Day 42
Population: Intent-to-treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | V565 | Placebo
Number analyzed (Participants) | 82 | 43
Participants | 29 | 16

2. Secondary Outcome: Number of Subjects Achieving Response to Therapy, Defined as Reduction in the CDAI Score and in Inflammatory Markers CRP or FCP at Day 42.
Description: Number of subjects achieving a ≥ 100-point reduction in CDAI score and a concomitant reduction of at least 50% in CRP or FCP at Day 42
  Crohn's Disease Activity Index (CDAI) is used to assess the symptoms of participants with Crohn's Disease. Scores generally range from 0 to 600, where clinical remission of Crohn's disease is defined as CDAI < 150, and very severe disease is defined as CDAI > 450.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | V565 | Placebo
Number analyzed (Participants) | 82 | 43
Participants | 20 | 9

3. Other Pre Specified Outcome: Number of Subjects With Improvement in Endoscopic Mucosal Appearance
Description: Subjects with a pre-treatment endoscopy Simple Endoscopic Score for Crohn's Disease (SES-CD) of at least 7 (4 if disease was confined to ileum) had a post-treatment endoscopy to evaluate changes in mucosal appearance. The central reader of the endoscopies, blinded to treatment and sequence, was asked to grade if video A was better or worse than video B. Pre- and post-treatment videos were randomly assigned to A and B. The endpoint is the number of subjects whose post-treatment endoscopy was better than their pre-treatment endoscopy.
Time Frame: Day 42
Population: Only those subjects who had a second endoscopy are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | V565 | Placebo
Number analyzed (Participants) | 32 | 10
Participants | 18 | 3

4. Other Pre Specified Outcome: Number of Subjects Achieving CRP Levels Within Normal Limits at Days 14 and 42
Description: The number of subjects who entered the study with an elevated CRP who had a CRP level within normal limits at Days 14 and 42.
  Normal levels defined as CRP less than or equal to 5mg/L
Time Frame: Days 14 and 42
Population: Patients were enrolled into the study based on either a baseline CRP measurement or a baseline FCP measurement. Only the subjects who entered the study based on their CRP measurement are included here.
Measure: Count of Participants; unit: Participants
Arm/Group | V565 | Placebo
Number analyzed (Participants) | 58 | 31
Participants | 11 | 4

5. Other Pre Specified Outcome: Number of Subjects Achieving FCP Levels Within Normal Limits at Day 14 and 42
Description: The number of subjects who entered the study with an elevated FCP who had an FCP level within normal limits at Days 14 and 42.
  Normal limits of FCP defined as less than or equal to 250µg/g
Time Frame: Days 14 and 42
Population: Patients were enrolled into the study based on either a baseline CRP measurement or a baseline FCP measurement. Only the subjects who entered the study based on their FCP measurement are included here.
Measure: Count of Participants; unit: Participants
Arm/Group | V565 | Placebo
Number analyzed (Participants) | 23 | 10
Participants | 7 | 3

ADVERSE EVENTS:
Time Frame: From Day 1 (first day of study medication) to Day 56 (14 days after last dose of study medication)
Arm/Group | V565 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/43
Serious Adverse Events (participants affected / at risk) | 3/82 | 2/43
Other Adverse Events (participants affected / at risk) | 30/82 | 16/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V565 (N=82) | Placebo (N=43)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Crohns Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) — Worsening of Crohn's Disease 7 days after the last dose of study medication
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V565 (N=82) | Placebo (N=43)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 4 (4)
Crohn's Disease (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (3) | 0 (0)
Pulpitis dental (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT02976129/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02976129/SAP_001.pdf